CLINICAL TRIAL: NCT00196573
Title: A Randomized Clinical Trial Comparing the Effectiveness of Subacromial Decompression (Acromioplasty) Versus Subacromial Bursectomy (no Acromioplasty) in the Arthroscopic Treatment of Patients With Rotator Cuff Tendinosis
Brief Title: Subacromial Decompression Versus Subacromial Bursectomy for Patients With Rotator Cuff Tendinosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Fowler Kennedy Sport Medicine Clinic (Other)
Responsible Party: Principal Investigator, Dianne Bryant, Associate Professor, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FKSMC-AOSSM-1; WillitsYIG1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Tendinosis; Shoulder Impingement Syndrome
Keywords: Rotator Cuff; Tendinosis; Impingement Syndrome; Partial Thickness Tears; Rotator Cuff Tendinosis; Partial Thickness Rotator Cuff Tears
MeSH Terms: conditions — Tendinopathy; Shoulder Impingement Syndrome; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (1):
- Shoulder bursectomy and acromioplasty (Active Comparator)
  Interventions: Procedure: Shoulder bursectomy alone

INTERVENTIONS:
Procedure: Shoulder bursectomy alone

SUMMARY:
The purpose of this study is to compare the effectiveness of arthroscopic subacromial decompression (acromioplasty) to arthroscopic subacromial bursectomy (no acromioplasty) in rotator cuff impingement syndrome. The investigators' hypothesis is that arthroscopic subacromial decompression provides no additional benefit, as evaluated with disease specific quality of life measures, compared to arthroscopic bursectomy.

DETAILED DESCRIPTION:
The most commonly performed surgical procedure to treat rotator cuff tendinosis, when no full-thickness tear exists, is subacromial decompression (acromioplasty). This procedure is based on the theory that primary acromial morphology, (an extrinsic cause), is the initiating factor leading to the dysfunction and eventual tearing of the rotator cuff.

Subacromial decompression involves surgical excision of the subacromial bursa, resection of the coracoacromial ligament, resection of the anteroinferior portion of the acromion, and resection of any osteophytes from the acromioclavicular joint that are thought to be contributing to impingement.

Several studies have indicated that the vast majority of partial-thickness tears are found on the articular surface of the rotator cuff which is not in keeping with the theory that rotator cuff impingement is primarily a result of acromion morphology.

Burkhart proposed that pathologic changes in the supraspinatus tendon occur primarily as a result of overuse and tension overload (an intrinsic factor), resulting in superior migration of the humeral head during active elevation.

Budoff et al., suggest that since the coracoacromial ligament stabilizes the rotator cuff to prevent uncontrolled superior migration of the humeral head, resection of the coracoacromial ligament during arthroscopic subacromial decompression may cause, in the long-term, additional proximal migration of the humeral head.

Arthroscopic bursectomy with debridement of rotator cuff tears alone, without acromioplasty, addresses the primary anatomical pathology and may offer similar success rates to subacromial decompression, without the risk of future instability caused by resection of the acromion and coracoacromial ligament.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stage II rotator cuff impingement syndrome defined as:

   * Pain referred to the anterior, lateral, or superior shoulder
   * Pain exacerbated by overhead and reaching activities
   * Positive Neer and/or Hawkins impingement signs
2. Failure of 6 months of conservative treatment. Failed conservative treatment will be defined as persistent pain and disability despite adequate non-operative management for 6 months. Non-operative management will be defined as:

   * Modification of activities
   * The use of analgesic and/or anti-inflammatory medication
   * Physiotherapy: Physiotherapy must have included the goal of regaining full range of motion, working towards normal kinematics through increased strength of the rotator cuff muscles. Patients should have obtained range of motion to 80% of the opposite shoulder (assuming this is normal) for each of: internal rotation, external rotation, and forward elevation. A physiotherapy program that involved massage, ultrasound, and/or heat only would not be considered adequate treatment for this study.
3. Patients willing to be followed on a regular basis
4. Patients 18 years of age and older

Exclusion Criteria:

1. Clinical evidence or history of major joint trauma, infection, surgery, glenohumeral arthritis, or instability.
2. Clinical evidence of internal impingement.
3. Patients with full-thickness rotator cuff tear as documented on advanced imaging or during surgery.
4. Patients with bursal surface tears as documented on advanced imaging or during surgery.
5. Patients who are found during surgery to have a partial-thickness tear greater than 50% of tendon thickness.
6. Patients with evidence of a lateral down sloping acromion.
7. Patients unfit for surgery
8. Patients unable to provide informed consent or adequately participate in this study due to a language barrier or psychiatric illness.
9. Patients with a major medical illness whose condition or treatment would affect their quality of life and, as such, affect the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2003-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario Rotator Cuff (WORC) index | Baseline, 2 & 6 weeks, 3, 6, 12, 18, 24 months
  a disease specific quality of life measure for rotator cuff disease evaluated pre-operatively and at all post-operative visits

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Willits, MD, FRCS(C), Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (6):
- Canada (6):
  - University of Calgary Sport Medicine Centre, Calgary, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Pan Am Medical and Surgical Centre, Winnipeg, Manitoba
  - Fowler Kennedy Sport Medicine Clinic, London, Ontario
  - Hand and Upper Limb Clinic, London, Ontario
  - Orthopaedic and Arthritic Hospital, Toronto, Ontario

REFERENCES:
- [Background] Altchek DW, Warren RF, Wickiewicz TL, Skyhar MJ, Ortiz G, Schwartz E. Arthroscopic acromioplasty. Technique and results. J Bone Joint Surg Am. 1990 Sep;72(8):1198-207. PMID 2398090
- [Background] Alvarez C, Kirkley A. The development of a disease specific quality of life measurement tool for rotator cuff disease. Presented at 23rd Clinical Seminar in Orthopaedic Surgery, London, Canada. May, 1995.
- [Background] Andrews JR, Broussard TS, Carson WG. Arthroscopy of the shoulder in the management of partial tears of the rotator cuff: a preliminary report. Arthroscopy. 1985;1(2):117-22. doi: 10.1016/s0749-8063(85)80041-4. PMID 4091915
- [Background] Banas MP, Miller RJ, Totterman S. Relationship between the lateral acromion angle and rotator cuff disease. J Shoulder Elbow Surg. 1995 Nov-Dec;4(6):454-61. doi: 10.1016/s1058-2746(05)80038-2. PMID 8665291
- [Background] Barrett WP, Franklin JL, Jackins SE, Wyss CR, Matsen FA 3rd. Total shoulder arthroplasty. J Bone Joint Surg Am. 1987 Jul;69(6):865-72. PMID 3597500
- [Background] Bassett RW, Cofield RH. Acute tears of the rotator cuff. The timing of surgical repair. Clin Orthop Relat Res. 1983 May;(175):18-24. PMID 6839586
- [Background] Bigliani LU, Levine WN. Subacromial impingement syndrome. J Bone Joint Surg Am. 1997 Dec;79(12):1854-68. No abstract available. PMID 9409800
- [Background] Bretzke CA, Crass JR, Craig EV, Feinberg SB. Ultrasonography of the rotator cuff. Normal and pathologic anatomy. Invest Radiol. 1985 May-Jun;20(3):311-5. doi: 10.1097/00004424-198505000-00015. PMID 3897119
- [Background] BROWN JT. Early assessment of supraspinatus tears; procaine infiltration as a guide to treatment. J Bone Joint Surg Br. 1949 Aug;31B(3):423-5. No abstract available. PMID 18142154
- [Background] Budoff JE, Nirschl RP, Guidi EJ. Debridement of partial-thickness tears of the rotator cuff without acromioplasty. Long-term follow-up and review of the literature. J Bone Joint Surg Am. 1998 May;80(5):733-48. doi: 10.2106/00004623-199805000-00016. No abstract available. PMID 9611036
- [Background] Burkhart SS. Arthroscopic debridement and decompression for selected rotator cuff tears. Clinical results, pathomechanics, and patient selection based on biomechanical parameters. Orthop Clin North Am. 1993 Jan;24(1):111-23. PMID 8421604
- [Background] Burkhead WZ. Symposium: the rotator Cuff: debridement versus repair - part I. Contemporary Orthopedics 31:262-271, 1995.
- [Background] Burkhead WZ. Symposium: the rotator Cuff: debridement versus repair - part II. Contemporary Orthopedics 31:313-326, 1995.
- [Background] Butters KP, Rockwood CA Jr. Office evaluation and management of the shoulder impingement syndrome. Orthop Clin North Am. 1988 Oct;19(4):755-65. PMID 3050719
- [Background] Cofield RH. Rotator cuff disease of the shoulder. J Bone Joint Surg Am. 1985 Jul;67(6):974-9. No abstract available. PMID 4019548
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Background] Coomes EN, Darling LG. Effects of local steroid injection for supraspinatus tears - Controlled Study. Annals of the rheumatic diseases 35: 943, 1976.
- [Background] Crass JR, Craig EV, Thompson RC, Feinberg SB. Ultrasonography of the rotator cuff: surgical correlation. J Clin Ultrasound. 1984 Oct;12(8):487-91. doi: 10.1002/jcu.1870120806. PMID 6436327
- [Background] Deutsch A, Altchek DW, Schwartz E, Otis JC, Warren RF. Radiologic measurement of superior displacement of the humeral head in the impingement syndrome. J Shoulder Elbow Surg. 1996 May-Jun;5(3):186-93. doi: 10.1016/s1058-2746(05)80004-7. PMID 8816337
- [Background] Ellman H. Arthroscopic subacromial decompression: A preliminary report. Ortop Trans 19:43, 1985.
- [Background] Ellman H. Arthroscopic subacromial decompression: analysis of one- to three-year results. Arthroscopy. 1987;3(3):173-81. doi: 10.1016/s0749-8063(87)80061-0. PMID 3675789
- [Background] Ellman H. Diagnosis and treatment of incomplete rotator cuff tears. Clin Orthop Relat Res. 1990 May;(254):64-74. PMID 2182260
- [Background] Ellman H, Hanker G, Bayer M. Repair of the rotator cuff. End-result study of factors influencing reconstruction. J Bone Joint Surg Am. 1986 Oct;68(8):1136-44. PMID 3771595
- [Background] Ellman H, Kay SP. Arthroscopic subacromial decompression 2-5 year results. Orthop Trans 13:239, 1989
- [Background] Esch JC. Arthroscopic subacromial decompression and postoperative management. Orthop Clin North Am. 1993 Jan;24(1):161-71. PMID 8421609
- [Background] Esch JC, Ozerkis LR, Helgager JA, Kane N, Lilliott N. Arthroscopic subacromial decompression: results according to the degree of rotator cuff tear. Arthroscopy. 1988;4(4):241-9. doi: 10.1016/s0749-8063(88)80038-0. PMID 3233112
- [Background] Fu FH, Harner CD, Klein AH. Shoulder impingement syndrome. A critical review. Clin Orthop Relat Res. 1991 Aug;(269):162-73. PMID 1864035
- [Background] Fukuda H, Hamada K, Yamanaka K. Pathology and pathogenesis of bursal-side rotator cuff tears viewed from en bloc histologic sections. Clin Orthop Relat Res. 1990 May;(254):75-80. PMID 2323150
- [Background] Gartsman GM. Arthroscopic treatment of rotator cuff disease. J Shoulder Elbow Surg. 1995 May-Jun;4(3):228-41. doi: 10.1016/s1058-2746(05)80056-4. PMID 7552682
- [Background] Gartsman GM. Arthroscopic acromioplasty for lesions of the rotator cuff. J Bone Joint Surg Am. 1990 Feb;72(2):169-80. PMID 2303503
- [Background] Gerber C, Terrier F, Ganz R. The role of the coracoid process in the chronic impingement syndrome. J Bone Joint Surg Br. 1985 Nov;67(5):703-8. doi: 10.1302/0301-620X.67B5.4055864.
- [Background] Hawkins RJ, Brock RM, Abrams JS, Hobeika P. Acromioplasty for impingement with an intact rotator cuff. J Bone Joint Surg Br. 1988 Nov;70(5):795-7. doi: 10.1302/0301-620X.70B5.3192582.
- [Background] Hawkins RJ, Kennedy JC. Impingement syndrome in athletes. Am J Sports Med. 1980 May-Jun;8(3):151-8. doi: 10.1177/036354658000800302. PMID 7377445
- [Background] Hodler J, Fretz CJ, Terrier F, Gerber C. Rotator cuff tears: correlation of sonographic and surgical findings. Radiology. 1988 Dec;169(3):791-4. doi: 10.1148/radiology.169.3.3055040.
- [Background] Iannotti JP (Ed). Rotator Cuff Disorders. American Academy of Orthopaedic Surgeons Monograph Series. Park Ridge, Illinois, 1991.
- [Background] Jobe FW, Kvitne RS, Giangarra CE. Shoulder pain in the overhand or throwing athlete. The relationship of anterior instability and rotator cuff impingement. Orthop Rev. 1989 Sep;18(9):963-75. PMID 2797861
- [Background] Kibler WB, Chandler TJ. Functional scapular instability in throwing athletes. American Orthopaedic Society for Sports Medicine 15th Annual Meeting. Traverse City, Michigan, June 19-22, 1989.
- [Background] Levy HJ, Gardner RD, Lemak LJ. Arthroscopic subacromial decompression in the treatment of full-thickness rotator cuff tears. Arthroscopy. 1991;7(1):8-13. doi: 10.1016/0749-8063(91)90071-5. PMID 2009126
- [Background] Mack LA, Matsen FA 3rd, Kilcoyne RF, Davies PK, Sickler ME. US evaluation of the rotator cuff. Radiology. 1985 Oct;157(1):205-9. doi: 10.1148/radiology.157.1.3898216.
- [Background] Matsen FA III, Arntz CT. Subacromial Impingement, in Rockwood CA Jr, Matsen FA II (eds): The Shoulder. Philadelphia, WB Saunders, 1990, pg 623-648.
- [Background] Montgomery TJ, Yerger B, Savoie FH. Management of full thickness tears of the rotator cuff: a comparison of arthroscopic debridement with open repair. Presented at the 8th annual Open Meeting of American Shoulder and Elbow Surgeons, Washington, DC, 1992.
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder: a preliminary report. J Bone Joint Surg Am. 1972 Jan;54(1):41-50. No abstract available. PMID 5054450
- [Background] Neer CS 2nd. Impingement lesions. Clin Orthop Relat Res. 1983 Mar;(173):70-7. No abstract available. PMID 6825348
- [Background] Neer CS 2nd, Craig EV, Fukuda H. Cuff-tear arthropathy. J Bone Joint Surg Am. 1983 Dec;65(9):1232-44. PMID 6654936
- [Background] Nirschl RP. Rotator cuff tendinitis: basic concepts of pathoetiology. Instr Course Lect. 1989;38:439-45. PMID 2649591
- [Background] Ogilvie-Harris DJ, Wiley AM. Arthroscopic surgery of the shoulder. A general appraisal. J Bone Joint Surg Br. 1986 Mar;68(2):201-7. doi: 10.1302/0301-620X.68B2.3958003.
- [Background] Ogilvie-Harris DJ, Wiley AM, Sattarian J. Failed acromioplasty for impingement syndrome. J Bone Joint Surg Br. 1990 Nov;72(6):1070-2. doi: 10.1302/0301-620X.72B6.2246291.
- [Background] Ozaki J, Fujimoto S, Nakagawa Y, Masuhara K, Tamai S. Tears of the rotator cuff of the shoulder associated with pathological changes in the acromion. A study in cadavera. J Bone Joint Surg Am. 1988 Sep;70(8):1224-30. PMID 3417708
- [Background] Paulos LE, Franklin JL. Arthroscopic shoulder decompression development and application. A five year experience. Am J Sports Med. 1990 May-Jun;18(3):235-44. doi: 10.1177/036354659001800303. PMID 2372071
- [Background] Post M, Cohen J. Impingement syndrome. A review of late stage II and early stage III lesions. Clin Orthop Relat Res. 1986 Jun;(207):126-32. PMID 3720075
- [Background] Rockwood CA, Burkhead WZ. Management of patients with massive rotator cuff defects by acromioplasty and rotator cuff debridement. Orthop Trans 12:190-191, 1988.
- [Background] Snyder SJ. Evaluation and treatment of the rotator cuff. Orthop Clin North Am. 1993 Jan;24(1):173-92. PMID 8421610
- [Background] Snyder SJ, Pachelli AF, Del Pizzo W, Friedman MJ, Ferkel RD, Pattee G. Partial thickness rotator cuff tears: results of arthroscopic treatment. Arthroscopy. 1991;7(1):1-7. doi: 10.1016/0749-8063(91)90070-e. PMID 2009105
- [Background] Soble MG, Kaye AD, Guay RC. Rotator cuff tear: clinical experience with sonographic detection. Radiology. 1989 Nov;173(2):319-21. doi: 10.1148/radiology.173.2.2678247.
- [Background] Speer KP, Lohnes J, Garrett WE Jr. Arthroscopic subacromial decompression: results in advanced impingement syndrome. Arthroscopy. 1991;7(3):291-6. doi: 10.1016/0749-8063(91)90130-p. PMID 1750939
- [Background] Steel RGD, Torrie JH. Principles of procedures of statistics. A biometric approach (2nd ed). McGraw-Hill Book Co. New York, NY, 1980.
- [Background] Watson MS. Classification of the painful arc syndromes. Bayley JI, Kessel L (eds). Shoulder Surgery. New York, NY, Springer-Verlag New York INC, 1982.
- [Background] Wiener SN, Seitz WH Jr. Sonography of the shoulder in patients with tears of the rotator cuff: accuracy and value for selecting surgical options. AJR Am J Roentgenol. 1993 Jan;160(1):103-7; discussion 109-10. doi: 10.2214/ajr.160.1.8416605.
- [Background] Wickiewicz, TL. Glenohumeral kinematics in a muscle fatigue model: a radiographic study. Orthop Trans 18:178-179, 1994.
- [Background] Williams GN, Gangel TJ, Arciero RA, Uhorchak JM, Taylor DC. Comparison of the Single Assessment Numeric Evaluation method and two shoulder rating scales. Outcomes measures after shoulder surgery. Am J Sports Med. 1999 Mar-Apr;27(2):214-21. doi: 10.1177/03635465990270021701. PMID 10102104
- [Background] Yamaguchi K, Flatow EL. Arthroscopic evaluation and treatment of the rotator cuff. Orthop Clin North Am. 1995 Oct;26(4):643-59. PMID 7566910
- [Background] Uhthoff HK, Hammond DI, Sarkar K, Hooper GJ, Papoff WJ. The role of the coracoacromial ligament in the impingement syndrome. A clinical, radiological and histological study. Int Orthop. 1988;12(2):97-104. doi: 10.1007/BF00266972. PMID 3410622
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720